CLINICAL TRIAL: NCT01049386
Title: Methods to Examine Intestinal Permeability Under Different Conditions
Brief Title: Intestinal Permeability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: R.F. Witkamp, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 8738
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-01

CONDITIONS: Intestinal Permeability
Keywords: intestinal permeability; health; sugar absorption; intestinal permeability examined in different men (lean vs obese) and different conditions (no breakfast and high-fat breakfast)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar absorption test (Active Comparator): In 150 mL of water four different sugars will be dissolved. Absorption will be calculated based on concentrations of sugars in 0-5 hours urine and 0-24 h collected urine.
  Interventions: Other: No intervention; Procedure: Sugar absorption test
- Sugar absorption test and high-fat breakfast (Experimental): In 150 mL of water four different sugars will be dissolved. Absorption will be calculated based on concentrations of sugars in 0-5 hours urine and 0-24 h collected urine. Subjects will eat a high-fat breakfast together with the sugar drink, to investigate the disturbance caused by fat in intestinal absorption.
  Interventions: Other: No intervention; Procedure: Sugar absorption test

INTERVENTIONS:
Other: No intervention — In obese and lean subjects the intestinal absorption will be examined under normal conditions with sugar drink, and when disturbed by a high-fat breakfast.
Procedure: Sugar absorption test — On one of the test days the subjects will consume a high-fat breakfast.

SUMMARY:
Rationale: Intestinal permeability of subjects can vary depending on their health status. It is therefore important to be able to measure and quantify intestinal permeability in a standardized way. Subjects with intestinal complaints (like irritable bowel disorder) or obese subjects have been found to have increased intestinal permeability. Different physiological conditions might affect intestinal permeability (IP) further.

In the clinic, sugar absorption tests and different blood and urine markers have been used to quantify IP. The sugars sucrose, mannitol, sucralose and lactulose are absorbed differently in the small or large intestines, resulting in different sugar levels in urine. This indicates the level of intestinal permeability and the location of increased permeability which is more or less permeable.

A high-fat meal could be used as a challenge test to increase IP in subjects even further. After a high fat meal, lipopolysaccharide (LPS) could be co-transported with chylomicrons. Small amounts of LPS co-transit with dietary fat from the gut after a high-fat meal, which thereby increases plasma LPS concentrations.

Because of the above mentioned reasons, it could be relevant to determine intestinal permeability and plasma LPS concentration after consumption of a high-fat diet.

Different methods will be used to determine the intestinal permeability in lean and obese men, under different conditions. New parameters, like intestinal (I) fatty acid binding protein (I-FABP), liver (L)-FABP, LPS and inflammatory markers will be measured and related to outcomes of tests, to examine the relation with intestinal permeability.

The association of IP with whole body electrical resistance will be examined, to determine usefulness of a candidate non-invasive method for IP investigation.

DETAILED DESCRIPTION:
Study design: The study is designed as a randomized, cross-over and open study.

Study population: 16 healthy, lean (BMI 20-25 kg.m-2) and obese (BMI 30-35 kg.m-2) male subjects will participate in the study, aged between 18-45 years.

Intervention: On two different test days eight lean and eight obese men will be supplied with a sugar drink to examine intestinal permeability under normal conditions and in combination with an oral fat load to examine intestinal permeability under stressed conditions.

Main study parameters/endpoints: Intestinal permeability will be examined with an absorption test using four different sugars (sucrose, mannitol, sucralose and lactulose). New markers of intestinal permeability, like I-FABP, L-FABP, LPS and inflammatory markers will be measured as well.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire (P8738 F02; in Dutch)
   * results of the pre-study laboratory tests
2. Males aged ≥ 18 and ≤ 45 years at Day 01 of the study
3. Body Mass Index (BMI): for the lean : ≥ 20 and ≤ 25 kg/m2; obese ≥ 30 and ≤ 35 kg/m2
4. Normal Dutch eating habits as assessed by P8738 F02
5. Voluntary participation
6. Having given written informed consent
7. Willing to comply with the study procedures
8. Appropriate veins for blood sampling/cannula insertion according to TNO
9. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
10. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

Subjects with one or more of the following characteristics will be excluded from participation:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 30-90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalator administration of substances
3. Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease or hypertension, stomach and intestinal complaints (and medication), pre-diabetes and Diabetes Mellitus
4. Having stomach and/or intestinal complaints after consumption of a high-fat meal
5. Usage of NSAIDs and/or acetylsalicylic acid (for example ibuprofen, diclofenac, naproxen or aspirin)
6. Smoking
7. Alcohol consumption ( > 28 units/week)
8. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
9. Reported slimming or medically prescribed diet
10. Recent blood donation (<1 month prior to the start of the study)
11. Not willing to give up blood donation during the study.
12. Personnel of TNO Quality of Life, their partner and their first and second degree relatives
13. Not having a general practitioner
14. Not willing to accept information transfer, concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
intestinal absorption (measured with the four sugar absorption test) | 24 hours

SECONDARY OUTCOMES:
Different biomarkers for intestinal absorption. | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: W J Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands